CLINICAL TRIAL: NCT01577186
Title: Symptomatic Remission and Social Function in Patients Treated With Paliperidone ER
Brief Title: Symptomatic Remission and Social Function in Participants Treated With Paliperidone Extended Release (ER)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015667; R076477SCH4035 (Other: Johnson & Johnson Taiwan Ltd); PAL-TWN-MA3 (Other: Johnson & Johnson Taiwan Ltd)
Record Dates: First submitted 2012-04-12; First posted 2012-04-13 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Extended Release
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone Extended Release (ER) (Experimental)
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — Participants will receive paliperidone ER tablet in flexible dose range of 3 to 12 milligram per day (mg/day) orally once daily up to Week 12 as per Investigator's discretion.

SUMMARY:
The purpose of this study is to explore the relationship between achieving symptomatic remission status by means of the 8 items of Positive and Negative Syndrome Scale (PANSS), and personal and social functioning by means of the Personal and Social Performance (PSP) scale in participants treated with flexibly dosed paliperidone ER.

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention), multicenter (when more than one hospital or medical school team work on a medical research study) and prospective (study following participants forward in time) 12-week study. Participants can be either in- or outpatients. The total study duration will be 12 weeks for each participant and will include following visits: Screening, Week 0, 4, 8, and 12 (end of treatment or early withdrawal). Throughout the study, participants will receive paliperidone ER in a flexible dosing range of 3 to 12 milligram per day (mg/day). Efficacy will primarily be evaluated by PANSS and PSP scale. Participants' safety will also be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria for schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self)
* Participant is drug naive or participant's previous treatment is considered unsuccessful due to one or more of the following reasons: lack of efficacy, lack of tolerability or safety, lack of compliance and/or other reasons
* Participants or their legally acceptable representatives had signed an informed consent document indicating that they understand the purpose of and procedures required for the study and were willing to participate in the study
* Women must be postmenopausal for at least 1 year, surgically sterile, abstinent, or, if sexually active, agree to practice an effective method of birth control before entry and throughout the study and must have a negative urine pregnancy test at screening

Exclusion Criteria:

* Participants with use of clozapine, paliperidone extended release (ER), any conventional depot neuroleptic or Risperdal CONSTA during the last 3 months
* Participants with serious unstable medical condition, including known clinically relevant laboratory abnormalities
* Participants with history of neuroleptic malignant syndrome (high fever, rigid muscles, shaking, confusion, sweating more than usual, increased heart rate or blood pressure, or muscle pain or weakness)
* Participants with known hypersensitivity to paliperidone ER or risperidone
* Participants with inability to swallow the whole study medication tablet with aid of water

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan Ltd Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone ER: Participants received paliperidone ER tablet in flexible dose range of 3 to 12 milligram per day orally once daily up to Week 12 as per Investigator's discretion.
Period: Overall Study
Arm/Group | Paliperidone ER
Started | 480
Completed | 350
Not Completed | 130
Not completed — Adverse Event | 23
Not completed — Death | 1
Not completed — Lost to Follow-up | 28
Not completed — Withdrawal by Subject | 35
Not completed — Insufficient Response | 18
Not completed — Ineligible to Continue | 15
Not completed — Non-Compliant | 8
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone ER
Number analyzed (Participants) | 480
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218
  Male | 262

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Symptomatic Remission by Means of Positive and Negative Syndrome Scale (PANSS)
Description: The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self). The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent), 2 (minimal), 3 (mild), 4 (moderate), 5 (moderately severe), 6 (severe) and 7 (extreme). The total score ranges from 30 to 210 and higher score indicates greater severity. Symptomatic remission was defined as achieving intensity level of mild or moderate on PANSS scale by all 8 items as the determinants for symptomatic remission: delusions, unusual thought content, hallucinatory behavior, conceptual disorganization, mannerisms/posturing, blunted affect, social withdrawal, lack of spontaneity.
Time Frame: End of study (Up to Week 12)
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Paliperidone Extended Release (ER): Participants received paliperidone ER tablet in flexible dose range of 3 to 12 milligram per day orally once daily up to Week 12.as per Investigator's discretion.
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 426
percentage of participants | 11.74 [8.84 to 15.18]

2. Secondary Outcome: Social Functioning Scale (SFS) Score
Description: The SFS is a 36-item scale designed to assess social functioning in schizophrenia. It assesses abilities and performance in seven areas: social engagement, interpersonal communication, activities of daily living, recreation, social activities, competence at independent living, and occupation/employment. Total score ranges from 1 to 100 where higher score indicates a more favorable health state.
Time Frame: End of study (Up to Week 12)
Population: ITT population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment. Here 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 374
units on a scale | 44.99 (19.05)

3. Primary Outcome: Percentage of Participants Achieving Improvement in Personal and Social Performance (PSP) Score by at Least One Category on PSP Scale
Description: The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty). Percentage of participants achieving improvement in PSP score by at least one category was reported.
Time Frame: End of study (Up to Week 12)
Population: ITT population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 426
percentage of participants | 47.42 [42.59 to 52.28]

4. Other Pre Specified Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 12
Description: The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent) to 7 (extreme). The total score ranges from 30 to 210 and higher score indicates greater severity.
Time Frame: Baseline, Week 12
Population: ITT population included all participants who received at least 1 dose of study drug and had at least one post-baseline assessment. Here, 'n' signifies those participants who were evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 426
units on a scale
  Baseline (n=426) | 89.88 (29.60)
  Change at Week 12 (n=350) | -16.07 (19.64)

5. Other Pre Specified Outcome: Change From Baseline in Total Personal and Social Performance (PSP) Score at Week 12
Description: The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty).
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 426
units on a scale
  Baseline (n=426) | 47.07 (16.34)
  Change at Week 12 (n=350) | 9.05 (12.55)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Paliperidone ER
Serious Adverse Events (participants affected / at risk) | 37/480
Other Adverse Events (participants affected / at risk) | 169/480
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER (N=480)
Supraventricular Tachycardia (Cardiac disorders) | 1
Pulmonary Tuberculosis (Infections and infestations) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Aggression (Psychiatric disorders) | 1
Alcohol Abuse (Psychiatric disorders) | 1
Completed Suicide (Psychiatric disorders) | 1
Drug Abuse (Psychiatric disorders) | 1
Hallucination, Auditory (Psychiatric disorders) | 2
Impulsive Behaviour (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Major Depression (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 27
Suicide Attempt (Psychiatric disorders) | 1
Scrotal Ulcer (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER (N=480)
Constipation (Gastrointestinal disorders) | 15
Nasopharyngitis (Infections and infestations) | 11
Upper Respiratory Tract Infection (Infections and infestations) | 32
Weight Increased (Investigations) | 14
Dizziness (Nervous system disorders) | 20
Extrapyramidal Disorder (Nervous system disorders) | 56
Headache (Nervous system disorders) | 10
Somnolence (Nervous system disorders) | 10
Tremor (Nervous system disorders) | 23
Anxiety (Psychiatric disorders) | 12
Insomnia (Psychiatric disorders) | 21

LIMITATIONS AND CAVEATS:
Some Adverse Events summaries were reported based on estimates due to the fact that they were not prepared in the original study report and the relevant definitions of the data elements were not available for these summaries to be regenerated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less